CLINICAL TRIAL: NCT06724822
Title: A Pilot Human Investigation of the Safety, Tolerability, Effectiveness of the Aqua Medical Circumferential RF Vapor (RFV) Ablation System for Duodenal Mucosal Repeat Ablation Treatment for the Management of Type-2 Diabetes Mellitus (STEAM T-2 DM Retreatment Study) in Patients Who Were Non-Responders to Initial Duodenal Mucosal Ablation Treatment
Brief Title: RF Vapor Ablation Retreatment of Duodenal Mucosa in Non-responders With Type-2 Diabetes Mellitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aqua Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-1023-SA
Record Dates: First submitted 2024-11-30; First posted 2024-12-09 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Study arm- RF Vapor Ablation arm (Experimental): This is a single arm study. All enrolled patients will be included in this arm
  Interventions: Device: RF Vapor Ablation

INTERVENTIONS:
Device: RF Vapor Ablation — RF Vapor ablation of the duodenum

SUMMARY:
The purpose of this study is to test the hypothesis that re-treatment of the duodenal mucosa with RF vapor ablation will result in improvement in glycemic parameters, without complications (bleeding/ stricture / perforation) among subjects who failed to show improvement after initial treatment of the duodenal mucosa with RF vapor ablation.

DETAILED DESCRIPTION:
The aims of the study are:

1. Evaluate the safety of the device and retreatment procedure based on the reported adverse events that occur.
2. Evaluate the effectiveness of the device and procedure by comparing change in HbA1c from baseline to 168 days post retreatment procedure.
3. Evaluate device tolerability based on pain scores reported by patients.

The subject population for this study are adults (18-65 years of age) with type-2 diabetes mellitus who have received initial RF vapor ablation of the duodenal mucosa and had improvement in HbA1C of <0.5% at their six month evaluation.

Twelve subjects, previously enrolled in the STEAM T2DM Pilot study did not show adequate (>0.5%) response to initial RF vapor ablation treatment of the duodenal mucosa.

Minimum study duration per subject is 6 months.

The study comprises of 5 phases:

Screening, Pre-procedure tests, RF Vapor ablation procedure, Post vapor ablation follow up, identification and long term follow up of responders.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects previously enrolled and treated in the STEAM T2DM Clinical study.
2. Subjects with improvement in HbA1c of ≤0.5% or with HbA1c of ≥ 7.5% at the 6-month visit while participating in the STEAM T2DM study.
3. Agrees to use an additional glucose-lowering treatment (e.g., liraglutide, other OAD except for glyburide), if recommended by the study Investigator in case of persistent hyperglycemia.
4. Able to comply with study requirements and understand and sign the Informed Consent Form
5. Compliance with STEAM T2DM clinical protocol

Exclusion Criteria:

1. Non-compliance with STEAM T2DM clinical protocol
2. Diagnosis of Type-1 Diabetes
3. History of diabetic ketoacidosis or hyperosmolar nonketotic coma.
4. Probable insulin production failure, defined as fasting C Peptide serum <1 ng/mL (333pmol/l).
5. Previous use of any types of insulin for >1 month (at any time, except for treatment of gestational diabetes).
6. Current use of injectable medications for diabetes (insulin, GLP-1RA).
7. Current use of glyburide, a sulfonylurea (SU) glucose-lowering drug for diabetes.
8. History of severe hypoglycemia (more than 1 severe hypoglycemic event, as defined by need for third-party assistance, in the last year).
9. Known autoimmune disease, including but not limited to celiac disease, duodenal Crohn disease or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other systemic autoimmune connective tissue disorder
10. Previous GI surgery that could limit treatment of the duodenum such as Billroth 2, Roux-en-Y gastric bypass, or other similar procedures or conditions. (Prior laparoscopic sleeve gastrectomy (LSG) will not be an exclusion)
11. History of chronic or acute pancreatitis.
12. History of diabetic gastroparesis.
13. Known active hepatitis or active liver disease.
14. Acute gastrointestinal illness in the previous 7 days.
15. Known history of severe irritable bowel syndrome, radiation enteritis or other inflammatory bowel disease, such as Crohn's disease.
16. Known history of a structural or functional disorder of the esophagus that may impede passage of the device through the gastrointestinal tract or increase risk of esophageal damage during an endoscopic procedure, including moderate-severe (Grade C or D) esophagitis, dysphagia due to achalasia or stricture/stenosis, esophageal varices, esophageal perforation, or any other disorder of the esophagus.
17. Upper gastrointestinal conditions such as active ulcers, polyps, varices, strictures, congenital or acquired duodenal telangiectasia
18. Current use of anticoagulation therapy (such as warfarin) that cannot be discontinued for 7 days before and 14 days after the procedure.
19. Current use of P2Y12 inhibitors (clopidogrel, prasugrel, ticagrelor) that cannot be discontinued for 14 days before and 14 days after the procedure.
20. Unable to discontinue non-steroidal anti-inflammatory drugs (NSAIDs) during treatment through 4 weeks following the procedure. Use of acetaminophen and low dose aspirin is allowed.
21. Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 12 weeks prior to the baseline visit.
22. Use of drugs known to affect GI motility (e.g. Metoclopramide)
23. Use of weight loss medications such as Sibutramine (e.g. Meridia), Orlistat (e.g. Xenical), Phentermine or over-the-counter weight loss medications (prescription medication)
24. Currently taking, or unable to stop taking dietary supplements or herbal agents, including vitamin C or multivitamins containing vitamin C at >500 mg per day, multivitamins containing biotin (vitamin B7), and supplements for hair, skin, and nail growth. Multivitamins not containing biotin are permitted.
25. Significant cardiovascular disease, including known history of valvular disease, or myocardial infarction, heart failure, transient ischemic attack, or stroke within 6 months prior to the Screening Visit.
26. Mean of 3 separate blood pressure measurements >180 mmHg (systolic) or >100 mmHg (diastolic).
27. Estimated glomerular filtration rate (eGFR) ≤ 60 ml/min/1.73m2 (estimated by MDRD).
28. Known immunocompromised status, including but not limited to individuals who have undergone organ transplantation, chemotherapy, or radiotherapy within the past 12 months, who have clinically significant leukopenia, who are positive for the human immunodeficiency virus (HIV) or whose immune status makes the participant a poor candidate for clinical trial participation in the opinion of the investigator.
29. Active illicit substance abuse or alcoholism (>2 drinks/day regularly)
30. Active malignancy within the last 5 years (excluding non-melanoma skin cancers)
31. Women breastfeeding
32. Participating in another ongoing clinical trial of an investigational drug or device.
33. Any other mental or physical condition which, in the opinion of the study investigator, makes the participant a poor candidate for clinical trial participation.
34. Critically ill or has a life expectancy <3 years
35. Use of heart pacemaker or other electronic device implants
36. General contraindications to deep or conscious sedation, general anesthesia, high risk as determined by anesthesiologist (e.g., ASA score 4 or higher), or contraindications to upper GI endoscopy.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint | 1 month
  Number of subjects with reported device or procedure related SAEs or UADEs.
Efficacy Endpoint | 168 days
  Change in HbA1c from baseline to 168 days post retreatment procedure
Tolerability Endpoint | 14 days
  Descriptive statistics on Visual Analogue Scale(VAS) pain scores
  Descriptive statistics on Visual Analogue Scale(VAS) pain scores
  Descriptive statistics on Visual Analogue Scale (VAS) pain scores

SECONDARY OUTCOMES:
Change in HbA1c at 84 days post retreatment procedure | 84 days
  Change in HbA1c at 84 days post retreatment procedure
Change in HbA1c over time | 168 days
  Change in HbA1c by visit over time
Change in FPG from baseline | 168 days
  Change in Fasting Plasma Glucose from baseline to 84 and 168 days post retreatment procedure
Change in FPG over time | 168 days
  Change in FPG change by visit over time (168 days post retreatment procedure)
Proportion of ablation-treated subjects with an improvement in HbA1c from baseline | 168 days
  Proportion of ablation-treated subjects with an HbA1c improvement from baseline at 168 days.
Change in HOMA-IR | 168 days
  Changes in HOMA-IR by visit over time (168 days post procedure).
Change in UACR | 168 days
  Change in UACR from baseline to 168 days post retreatment procedure
Change in ALT | 168 days
  Change in ALT from baseline to 168 days post retreatment procedure.
Change in AST | 168 days
  Change in AST from baseline to 168 days post retreatment procedure.

OTHER OUTCOMES:
Long term follow up endpoints among responders: Change in HbA1c | 2 years
  Change in HbA1c over time among responders
Long term follow up endpoints among responders: Change in FPG | 2 years
  Change in FPG by visit over time among responders
Long term follow up endpoints among responders: Proportion of responders | 168 days
  Proportion of subjects that show improvement at 6 months post retreatment
Long term follow up endpoints among responders: Change in HOMA-IR | 2 years
  Changes in HOMA-IR by visit over time
Long term follow up endpoints among responders: Change in UACR | 2 years
  Change in UACR by visit over time

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Rodriguez, MD, Principal Investigator — Clinica Colonial, Santiago, Chile
Locations (1):
- Clinica Colonial, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No